CLINICAL TRIAL: NCT01087112
Title: A Follow-up Study of a Randomized Controlled Trial of Mother-Infant Psychoanalytic Treatment and Treatment As Usual at Child Health Centres
Brief Title: Mother-Infant Psychoanalysis Project of Stockholm (MIPPS)- Follow-up at 4½ Years
Acronym: MIPPS-02
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Björn Salomonsson, Dept. of Woman and Child Health, Child and Adolescent Psychiatry Unit, Karolinska Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIPPS-02
Record Dates: First submitted 2009-12-29; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2009-12

CONDITIONS: Mother-child Relationship Disturbances
Keywords: MIP; RCT; postnatal depression; Mother-child relationship
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child Health Centre care (Active Comparator): TAU involved scheduled health visitor calls at the local Child Health Centre (CHC), with paediatric checkups at 2 and 6 months of age. The health visitor is encouraged to promote attachment and to detect postnatal depressions. Mothers may be offered parental groups, infant massage or guidance promoting interaction, as well as appointments with a paediatrician or a child psychiatric psychologist. Additional treatment was initiated in 1/3 of the cases. This was registered at the end-point interview.
  Interventions: Behavioral: Child Health Centre care
- Mother-Infant Psychoanalytic tmt (Experimental): MIP (Norman, 2001; 2004) is a psychoanalytic method adapted to the requirements of the infant as analysand in the presence of his mother. The analyst strives to recruit the baby for an emotional interchange, though this does not imply any belief that the infant understands verbal communication. The analyst addresses the baby to help him liberate emotions consolidated in symptoms such as screaming, avoiding maternal eye contact, and breast refusal. The analyst takes great care in enrolling the participant mother. This is to enhance her understanding of the baby's predicament and the nature of their relation, as well as giving her all space needed to vent her own frustration, depression and anxiety.
  Interventions: Behavioral: Mother-Infant Psychoanalytic tmt

INTERVENTIONS:
Behavioral: Mother-Infant Psychoanalytic tmt — Psychoanalytic sessions with mother and infant, at a median of 23 sessions 2 times weekly.
  Other Names: MIP
  Arms: Mother-Infant Psychoanalytic tmt
Behavioral: Child Health Centre care — Nurse calls at Child Health Centres (CHC), with regular paediatric checkups. The nurse was encouraged to promote attachment and to detect postnatal depressions. Appointments with a psychiatrist or therapist or child psychiatric psychologist was initiated in 1/3 of the cases. This was registered at the end-point interview.
  Other Names: CHCC
  Arms: Child Health Centre care

SUMMARY:
An RCT comparing mother-infant psychoanalytic treatment (MIP) with Child Health Centre care in cases of mother-infant relationship disturbances was performed on 80 cases in Stockholm 2005-2008. The infants were < 18 months at interview #1. At 6 months follow-ups, significant effects were shown in favour of MIP on maternal sensitivity (EAS), depression (EPDS), and relationship qualities PIR-GAS). This study will evaluate effects at a child age of 4½ years; to evaluate the longterm effects of MIP and CHild Health Centre care, and to better validate results on children who now have reached an age where they can participate more actively in evaluations.

DETAILED DESCRIPTION:
DESIGN

The 71 dyads remaining from the MIPPS-01 study will be interviewed when the children have reached 4½ years, in order to evaluate the long-term intervention effects of MIP treatments delivered by psychoanalysts at the Infant Reception Service of the Swedish Psychoanalytic Society and of the usual treatments of infants and children in Sweden implying contact with nurses at Child Health Centres.

INSTRUMENTS

Mother-report questionnaires; the Ages and Stages Questionnaire:Social-Emotional (ASQ:SE; Squires et al., 2002), the Edinburgh Postnatal Depression Scale (EPDS; Cox et al., 1987), the Swedish Parental Questionnaire (SPSQ; Östberg et al., 1997) and the Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997).

Independently rated video-taped mother-child interactions: the Emotional Availability Scale (EAS; Biringen, 1998).

Assessment of the general functioning of the child : Children's Global Assessment Scale (Shaffer et al 1983).

Assessment of the child's cognitive functioning: Wechsler Preschool and Primary Scale of Intelligence (WPPSI, Wechsler, 2005).

Assessment of the child's social and emotional functioning: Story Stem Attachment Profile (SSAP, Hodges et al., 2003). Machover Draw-a-Person Test (Blomberg & Cleve, 1997)

ELIGIBILITY:
Inclusion Criteria:

* The mother expressed significant concerns about one or more of the following domains: herself as a mother, her infant's well-being, or the mother-baby relationship (this was operationalized as a score < 80 ("perturbed relation") on the PIR-GAS or, alternatively, > 2.5 on the SPSQ).
* Infant of any gender, age below 18 months.
* Duration of worries exceeding two weeks.
* Domicile in Stockholm.
* Reasonable mastery of Swedish.

Exclusion Criteria:

* Maternal psychosis according to DSM-IV, to an extent precluding collaboration.
* Substance dependence according to DSM-IV, to an extent precluding collaboration.

Ages: 54 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Child functioning: Children's Global Assessment Scale | At followup interview
Maternal depression: Edinburgh Postnatal Depression Scale | At followup interview

SECONDARY OUTCOMES:
Maternal distress: Symptom Check List - 90 | At followup interview
Maternal stress: Swedish Parental Stress Questionnaire | At followup interview
Child functioning: Ages and Stages Questionnaire:Social Emotional | At followup interview
Child functioning: Strengths and Difficulties Questionnaire | At followup interview
Child cognitive functioning: Wechsler's Preschool and Primary Scales of Intelligence | At followup interview
Child's social and emotional functioning: Story Stem Attachment Profile | At followup interview
Child's social and emotional functioning: Machover Draw-a-Person test | At followup interview

CONTACTS AND LOCATIONS:
Overall Officials: Björn Salomonsson, MD, Principal Investigator — Department of Women's and Children's Health, Child and Adolescent Psychiatry Unit, Karolinska Institutet; Majlis Winberg Salomonsson, M.Sci.Psych., Principal Investigator — Department of Women's and Children's Health, Child and Adolescent Psychiatry Unit, Karolinska Institutet
Locations (1):
- Department of Women's and Children's Health, Child and Adolescent Psychiatry Unit, Karolinska Institutet, Stockholm, Sweden